CLINICAL TRIAL: NCT03978273
Title: Effects of Real-Time Feedback Assisted Self-Correction on the Posture of Scoliotic Patients: A Prospective, Monocentric, Randomized With Stratification on the Type of Scoliosis, Comparative and Open-label Study
Brief Title: Effects of Real-Time Feedback Assisted Self-Correction on the Posture of Scoliotic Patients
Acronym: COVIRSCOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network); University Grenoble Alps (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC18.053
Record Dates: First submitted 2019-05-15; First posted 2019-06-07 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Idiopathic Scoliosis
Keywords: Vertebral column; Rehabilitation; Virtual-brace; Posture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Night-time brace + virtual-brace (Experimental): Patients are conventionally treated with night-time brace. Additionally, they use the new developped virtual-brace (MD).
  Interventions: Device: Night-time brace + virtual-brace
- Night-time brace only (Active Comparator): Patients are conventionally treated with night-time brace only.
  Interventions: Other: Night-time brace only

INTERVENTIONS:
Device: Night-time brace + virtual-brace — Patients will receive conventional treatment : wearing a night-time brace every night during 6 months.
  Additionally :
  * They will perform 5 sessions of postural rehabilitation exercises per week (each of 30 minutes) with the virtual-brace (MD).
  * They will have also follow up consultations with a physiotherapist every 21 days, to evaluate treatment observance and to adapt postural exercises according to the results and difficulties encountered.
  Conventional 3D motion capture Analysis (different trunk tasks and walk) will be performed to evaluate evolution of postural parameters at D0, D90 and D180.
  Arms: Night-time brace + virtual-brace
Other: Night-time brace only — Patients will receive conventional treatment : wearing a night-time brace every night during 6 months.
  Conventional 3D motion capture Analysis (different trunk tasks and walk) will be performed to evaluate evolution of postural parameters at D0, D90 and D180.
  Arms: Night-time brace only

SUMMARY:
Scoliosis is a progressive three-dimensional deformation of the spine during growth, with a prevalence of 80% in girls.

The treatments currently used are surgery and rigid brace, which aim to stabilize scoliosis evolution. The place of rehabilitation is disputed because the methods are multiple, non-standardized and the sessions are infrequent.

In a previous study (MOUVSCO, NTC02134704), researchers have identified systematic postural abnormalities in patients with scoliosis, and developped a virtual-brace (medical device, MD) to allow real-time self-correction of the trunk position.

The aim of the present study is to evaluate for the first time the efficacy of the virtual-brace on the correction of the posture of scoliotic patients.

The hypothesis is that intensified rehabilitation with the virtual-brace will improve pathological postures related to scoliosis.

DETAILED DESCRIPTION:
The present study is the first evaluation of the efficacy of the virtual-brace on scoliotic patients.

The efficacy of rehabilitation will be estimate on the correction of the posture of scoliosis patients over 6 months by comparing 2 groups: a control group of patients conventionally treated with a night-time brace (G0 group_conventional) and an experimental group of patients wearing a night-time brace, doing postural rehabilitation exercises with the virtual brace and follow-up visits with a physiotherapist (G1 group_virtual-brace).

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic scoliosis (left lumbar or right thoracic),
* Patients with moderate scoliosis: Cobb angle assessed on the last radiography between 20 ° and 35 °,
* Patients requiring the wearing of a rigid night-time brace,
* Patients having a home computer,
* Patients affiliated to social security or similarly regime,
* Patients who gave their consent to participate in the study,
* Patients whose 2 parents have signed the informed consent

Exclusion Criteria:

* Patients with an unstabilized medical problem,
* Patients with known allergy to elastane,
* Patients with sensitivity to dizziness,
* Patients with pacemaker,
* Patients with implanted cardiac defibrillator,
* Patients with cochlear implant,
* Patients carrying a non-removable metal element,
* Protected patient concerned by articles L1121-5 and L1121-6 of the Public Health Code,
* Patients whose parents are protected by article L1121-8 of the Public Health Code

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Medio-lateral displacement during lateral inclination of scoliosis patients in the group with rehabilitation enriched by the virtual brace (group G1) compared with the reference treatment (group G0) at D180. | 6 months
  Difference between D180 and D0 of the medio-lateral displacement of the pressure center during the lateral inclination in both groups G0 and G1. This parameter is evaluated during the conventional 3D motion capture analysis.

SECONDARY OUTCOMES:
Quantification of kinematic, postural and electromyographic anomalies during trunk tilting and rotation (for both groups G0 and G1). | 6 months
  Conventional 3D motion capture analysis with surface ElectroMyoGram (EMG) pattern's at D0, D90 and D180.
Quantification of the quality of life evaluated with the Scoliosis Research Society Patient questionnaire (SRS-22), for both groups G0 and G1. | 6 months
  Difference in the result of the SRS-22 questionnaire between D180 and D0. SRS-22 is a self-reported questionnaire assessing self-image, function, pain, mental health, and satisfaction with care with score range from 1 to 5 (1=worst and 5= best) for each 22 questions. The global score is the mean score of all questions.
Quantification of kinematic feedback provided by the virtual-brace and their deviation from the prescription (only for group G1) | 6 months
  Time course of the angular data of the trunk relative to the pelvis provided by the virtual brace, versus the prescribed exercises (evaluated every 3 weeks during the visit to the physiotherapist)
Treatment compliance for the rigid-brace (for both group G1 and G0) | 6 months
  Compliance with the wearing of the rigid brace reported in the patient follow-up logbook.
Treatment compliance for the virtual-brace (only for group G1) | 6 months
  Only for group G1 : effective rehabilitation time collected from the virtual brace's log files.
Quantification of electroencephalogram (EEG) modifications during postural and walk initiation tasks (for both groups G0 and G1). | 6 months
  Conventional 3D motion capture analysis with EEG records at D0, D90 and D180.
Exploratory Objective : Descriptive analysis by group of all parameters related to postural disorders recorded during Conventional 3D motion capture analysis with EMG, EEG. | 6 months
  Set of variables related to the severity of the postural disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Aurelien COURVOISIER, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No